CLINICAL TRIAL: NCT03104010
Title: A Non-inferiority Phase 2 Study to Evaluate the Safety and Efficacy of PEG-rhGH in the Treatment of Adult Growth Hormone Deficiency (AGHD)
Brief Title: A Non-inferiority Phase 2 Study to Evaluate the Safety and Efficacy of PEG-rhGH in the Treatment of AGHD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Peking Union Medical College Hospital (Other); Peking University First Hospital (Other); Hebei General Hospital (Other); The Second Hospital of Hebei Medical University (Other); Qilu Hospital of Shandong University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); The First Affiliated Hospital of Soochow University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Chongqing Three Gorges Central Hospital (Other); West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 034 CT
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-rhGH-1 (Experimental): Pegylated recombinant human growth hormone injection, 12IU/2.0mg/1.0ml/bottle. The first stage, 1-2mg/2-4mg, subcutaneous injection,weekly, 26 weeks.
  Interventions: Drug: Somatropin Injection
- PEG-rhGH-2 (Experimental): Pegylated recombinant human growth hormone injection, 12IU/2.0mg/1.0ml/bottle. The second stage (extension period study), maximum ≤4mg/w (24IU/w), 52 weeks.
  Interventions: Drug: Somatropin Injection

INTERVENTIONS:
Drug: Somatropin Injection — Recombinant human growth hormone injection, 15IU/5mg/3ml/bottle. The first stage , 0.17mg/d(0.5IU/d), subcutaneous injection ,daily, 26weeks. The second stage(extension period study), 0.17mg/d(0.5IU/d), maximum ≤0.68mg/d (2IU/w),52 weeks.
  Other Names: Recombinant human growth hormone injection

SUMMARY:
This study aims to explore the optimal dose of PEG-rhGH injection in the treatment of AGHD, preliminarily evaluate its safety and efficacy, to provide scientific and reliable evidence for the medication dosage in Phase 2 clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Before the treatment, the subject should be diagnosed as AGHD based on medical history, clinical symptoms, vital signs, insulin tolerance test and imagological examinations.

  * The subject is diagnosed as GHD during childhood and remains as GHD in adulthood, and the linear growth has completed: bone age (BA) ≥18 years old; or the AGHD patient who experiences paroxysm after 18 years old: such as patients who have experienced pituitary surgeries (2 years after pituitary adenoma surgery, 5 years after craniopharyngioma surgery and 12 months after other pituitary surgeries), traumatic brain injury (TBI), Sheehan syndrome, and etc..
  * The plasma GH concentration peak is <5ng/ml in insulin tolerance test (ITT) (it's unnecessary to conduct ITT in the following conditions: anterior pituitary dysfunction, pituitary hormone deficiency (more than 3 hormones) and serum IGF-1 level below lower limit of normal value: i.e. -2 SD).
* Age: 18-60 years old.
* Patients with no history of GH treatment for more than one year.
* Body mass index (BMI): 18.5 kg/m2≤BMI≤30kg/m2.
* When there is other hormones deficiency (such as glucocorticoids, thyroid hormones and sex steroids), the subject should have received other hormone replacement therapies and the therapeutic dose shall be stable within 3 months before the enrolment.
* The subject agrees to cooperate and complete the concerted trial procedures such as follow-ups, treatment plan and laboratory examinations, and sign the written informed consent.

Exclusion Criteria:

* Patients with serious heart diseases, including NYHA III or above, serious arrhythmia, unstable angina pectoris or myocardial infarction within the latest 6 months.
* Patients with a history of ischemic cerebrovascular disease, febrile convulsion and epilepsy seizures.
* Patients with carpal tunnel syndrome.
* Patients with poor hypertension control (systolic pressure>140mmHg or diastolic pressure >90mmHg under treatment).
* Patients with previous or present history of malignant tumor: two or more direct relatives within three generations have previous or present history of tumor.
* Patients undergoing anti-depressive therapy, immunosuppressive therapy, chemotherapy and radiotherapy (or with a history of radiotherapy).
* Patients who have ever taken antiobesity drug within the latest 3 months.
* Patients with serious infection.
* Patients with consciousness disorders and mental diseases.
* Subjects with impaired glucose regulation (IGR) (impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT) ) or diabetes; patients with a family history of diabetes (direct relatives).
* Subjects with abnormal liver and kidney functions (ALT > 2 times of upper limit of normal value; eGFR calculated by MDRD formula <60).
* Subjects positive for anti-HBc, HBsAg or HBeAg in Hepatitis B virus tests.
* Subjects with highly allergic constitution or allergy to proteins or investigational productorits excipient in this study.
* Subjects who took part in other clinical trials within 3 months.
* Patients with other mental or physical deficiencies that influence the evaluation of investigational product.
* Pregnant or lactating women; females planning to get pregnant within one year.
* Subjects whose tumor markers exceed the upper limit of normal range and the re-examination result is still high.
* Other conditions which is unsuitable for the study in the opinion of the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Fat mass change | 52 weeks
  Change from baseline in fat mass (torso) (FM): FM at the end of treatment minus the baseline value

SECONDARY OUTCOMES:
Lean body mass change | 52 weeks
  Change from baseline in lean body mass (LBM): LBM at the end of treatment minus the baseline value
Blood lipid change | 52 weeks
  Change from baseline in blood lipid: blood lipid at the end of treatment minus the baseline value
Waist circumference change | 52 weeks
  Change from baseline in waist circumference: waist circumference at the end of treatment minus the baseline value
Percentage of body fat change | 52 weeks
  Change from baseline in the percentage of body fat: TBF at the end of treatment minus the baseline value
Cardiac function change | 52 weeks
  Change from baseline in cardiac function: ejection fraction at the end of treatment minus the baseline value
Cardiac structure change | 52 weeks
  Change from baseline in cardiac structure: left ventricular mass at the end of treatment minus the baselines value
IGF-1 change | 52 weeks
  Changes from baseline in IGF-1: IGF-1 SDS at the end of treatment minus the baseline value
Grip change | 52 weeks
  Changes from baseline in grip: grip at the end of treatment minus the baseline value, the method of assessment is measurement.
Quality of life change | 52 weeks
  Changes from baseline in quality of life (QOL): changes in QOL scores before and after treatment
Waist-hip ratio change | 52 weeks
  Changes from baseline in waist-hip ratio: changes of waist-hip ratio before and after treatment
Cardiac structure change | 52 weeks
  Change from baseline in cardiac structure: carotid intima media thickness at the end of treatment minus the baselines value

CONTACTS AND LOCATIONS:
Overall Officials: Hui Pan, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (9):
- China (9):
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Heibei General Hospital, Shijiazhuang, Hebei
  - The Affiliated hospital of soochow University, Suzhou, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University school of medicine, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - Chongqing Three Gorges Central Hospital, Chongqing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing